CLINICAL TRIAL: NCT06682260
Title: Impact of Nitroglycerin-induced Vasodilation on Stroke Volume and Diuretic Response in Acute Heart Failure: a Protocol for a Mechanistic Trial
Brief Title: Evaluating the Effects of Nitroglycerin on Heart Function and Urinary Output in Patients with Acute Heart Failure
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Copenhagen University Hospital, Hvidovre (Other)
Responsible Party: Principal Investigator, Frederik Lau, Medical Doctor, Copenhagen University Hospital, Hvidovre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Nitro-vers.1.1.
Record Dates: First submitted 2024-11-07; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Acute Heart Failure (AHF)
Keywords: Acute heart failure; Vasodilation; Nitroglycerin; Hemodynamics; Stroke volume; Cardiac function
MeSH Terms: conditions — Aneurysm | interventions — Nitroglycerin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Nitroglycerin (Experimental): Infusion of intravenous nitroglycerin titrated towards a vasodilatory state which we predefined as a 20-30% decrease in mean arterial pressure (MAP) for 1.5 hours followed by a phase of 1.5 hours with no vasodilation.
  Interventions: Drug: Nitroglycerin (NTG)

INTERVENTIONS:
Drug: Nitroglycerin (NTG) — Infusion of intravenous nitroglycerin beginning at 2 microgram/kg/min (2 ml/hour) and titrated with the aim of a MAP reduction of 20-30%. Infusion rate will not be increased after the first 30 minutes and is limited to 0.1 µg/kg/min to 5 µg/kg/min.

SUMMARY:
This study aims to understand how nitroglycerin affects patients with acute heart failure, a condition where the heart struggles to pump blood effectively, leading to fluid buildup and breathing difficulties. Nitroglycerin relaxes blood vessels to ease the heart's workload and may help reduce fluid buildup. The investigators hypothesize that nitroglycerin can increase blood flow from the heart and promote urine production, which may reduce congestion in AHF patients. By studying heart function, blood volume, and fluid levels during treatment, the goal is to identify which patients may benefit most from nitroglycerin therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Clinical diagnosis of AHF requiring hospitalization
* Systolic blood pressure ≥85 mmHg
* Echocardiographic signs of cardiac dysfunction, by at least one of

  * Left ventricular ejection fraction ≤45%
  * Abnormal left ventricular filling with dilatation of the left atrium
  * Elevated filling pressures (systolic pulmonary artery pressure>30, dilated vena cava inferior or E/é>10)
  * Significant left-sided heart valve disease

Exclusion Criteria:

* Ongoing ventricular taky- or brady-arrythmias or supraventricular arrhythmias with heart rate > 180 or < 40 bpm.
* Retinopathy or intraocular lens implantation (contraindication to Valsalva maneuver)
* Recent myocardial infarction or thromboembolic events.
* Intake of sildenafil or vardenafil withing 24 h and tadalafil within 48 h.
* Absolute contraindication for vasodilation using nitroglycerin as assessed by treating physician
* Intravenous administration of furosemide within 2 hours of baseline measurements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Stroke volume | From initiation of nitroglycerin infusion at time zero until study termination at 180 minutes.
  Change in stroke volume (obtained from LiDCO) from baseline through vasodilation period.

SECONDARY OUTCOMES:
Cumulated urinary output (mL) | From time zero until study termination at 180 minutes.
  Measurement of cumulated urinary output after placement of a transurethral catheter.
Mean arterial blood pressure | From time zero throughout the study period until termination at time 180 minutes.
Heart rate | From time zero throughout the study period until termination at time 180 minutes.
Cardiac output | At baseline and at timepoints 90 minutes and 180 minutes.
  Measured by echocardiography.
Peripheral perfusion index | From time zero throughout the study period until termination at time 180 minutes.
  As obtained by photoplethysmography, where a higher numerical value may indicate better peripheral tissue perfusion.
Systemic vascular resistance | From time zero throughout the study period until termination at time 180 minutes.
  [SVR=(MAP-RAP)×80/CO]

IPD SHARING:
Plan to Share IPD: No
It is not possible for data to be shared due to legal reasons.